CLINICAL TRIAL: NCT01550965
Title: An Open-Label Multicenter Study to Evaluate the Impact of Adalimumab on Quality of Life, Health Care Utilization and Costs of Ulcerative Colitis Subjects in the Usual Clinical Practice Setting
Brief Title: A Study to Evaluate the Impact of Adalimumab on Quality of Life, Health Care Utilization and Costs of Ulcerative Colitis Subjects in the Usual Clinical Practice Setting
Acronym: InspirAda
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M13-045; 2011-002411-29 (EudraCT Number)
Record Dates: First submitted 2012-03-08; First posted 2012-03-12 (Estimated); Results first posted 2016-11-01 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2016-05

CONDITIONS: Ulcerative Colitis
Keywords: Quality of Life; Costs of Ulcerative Colitis; Health Care Utilization
MeSH Terms: conditions — Colitis, Ulcerative; Patient Acceptance of Health Care | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Participants Receiving Adalimumab (Experimental): Adults with active UC who had failed conventional therapy received Adalimumab 160 mg at Baseline Visit, 80 mg at Week 2 Visit, and 40 mg every other week (EOW) starting at Week 4. Non-responders to adalimumab were to be discontinued from treatment at Week 8. After Week 8, dose escalation to 40 mg weekly was allowed for flare or non-response.
  Interventions: Biological: Adalimumab

INTERVENTIONS:
Biological: Adalimumab — Adalimumab pre-filled syringe, administered by subcutaneous injection
  Other Names: ABT-D2E7; Humira®

SUMMARY:
This study evaluated the quality of life (QOL) and economic impact of adalimumab treatment in participants with ulcerative colitis (UC).

DETAILED DESCRIPTION:
This was a single arm, open-label, multicenter study. The primary objectives were to study the effect of adalimumab on QOL (as measured by Short Inflammatory Bowel Disease Questionnaire (SIBDQ)), the utilization of health care resources, and the costs of care for subjects with UC who were treated with adalimumab in the usual clinical practice setting. The secondary objectives were to further assess the effect of adalimumab on disease activity and to collect additional safety data in subjects with UC.

ELIGIBILITY:
Inclusion Criteria:

1. Participants had to be a male or female between the ages of 18 and 75 years old at the time of the Screening Visit.
2. Participants who had a diagnosis of ulcerative colitis (UC) greater than 90 days prior to baseline (week 0) and failed conventional treatment.
3. Participants diagnosis of active UC was confirmed by a colonoscopy with biopsy or flexible sigmoidoscopy with biopsy.
4. Participants who had active UC with a Physicians Global Assessment (PGA) score of 2 or 3 and Short Inflammatory Bowel Disease Questionnaire (SIBDQ) ≤ 45 at baseline (week 0).
5. Concurrent therapy was required for participants who were previously treated with corticosteroids or immunosuppressants (azathioprine (AZA) or 6-mercaptopurine (6-MP)) and, in the judgment of the investigator, had failed to respond to or could not tolerate their treatment. Participants had to be on a concurrent treatment with at least one of the following (oral corticosteroids or immunosuppressants or both as defined below):

   * Stable oral corticosteroid dose (prednisone ≥ 20 mg/day or equivalent) for at least 14 days prior to baseline, or
   * Stable oral corticosteroid dose (prednisone < 20 mg/day) for at least 21 days prior to baseline, and/or
   * At least a consecutive 12 weeks (84 days) course of AZA or 6-MP prior to baseline.

Exclusion Criteria:

1. Participants who had a history of subtotal colectomy with ileorectostomy or colectomy with ileoanal pouch, Kock pouch, or ileostomy for UC or planned bowel surgery.
2. Participants received previous treatment with adalimumab or previous participation in an adalimumab clinical study.
3. Participants who had previously used infliximab or any anti- tumor necrosis factor (TNF) agent within 56 days of baseline (week 0).
4. Participants who had previously used infliximab or any anti-TNF agent and had not clinically responded at any time ("primary non-responder") unless they experienced a treatment limiting reaction.
5. Participants who had received cyclosporine, tacrolimus, or mycophenolate mofetil within 30 days of baseline (week 0).
6. Participants who had received intravenous (IV) corticosteroids within 14 days of Screening or during the screening period.
7. Participants who had a current diagnosis of fulminant colitis and/or toxic megacolon.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 463 (Actual)
Dates: Start 2012-05; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Medich, Study Director — AbbVie

REFERENCES:
- [Result] Travis S, Feagan BG, Peyrin-Biroulet L, Panaccione R, Danese S, Lazar A, Robinson AM, Petersson J, Pappalardo BL, Bereswill M, Chen N, Wang S, Skup M, Thakkar RB, Chao J. Effect of Adalimumab on Clinical Outcomes and Health-related Quality of Life Among Patients With Ulcerative Colitis in a Clinical Practice Setting: Results From InspirADA. J Crohns Colitis. 2017 Oct 27;11(11):1317-1325. doi: 10.1093/ecco-jcc/jjx093. PMID 28981846
- See also: Related Info — http://www.rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 463 participants were enrolled: 461 in the intent to treat (ITT) population were analyzed for efficacy (excluding 2 due to lack of post-baseline measurement data); 463 were analyzed for safety (participants who had received at least one dose of study drug).
Groups:
- Participants Receiving Adalimumab: Adults with active ulcerative colitis (UC) who had failed conventional therapy received Adalimumab 160 mg at Baseline Visit, 80 mg at Week 2 Visit, and 40 mg every other week (EOW) starting at Week 4. Non-responders to adalimumab were to be discontinued from treatment at Week 8. After Week 8, dose escalation to 40 mg weekly was allowed for flare or non-response.
Period: Overall Study
Arm/Group | Participants Receiving Adalimumab
Started | 463
Completed | 353
Not Completed | 110
Not completed — Adverse Event | 26
Not completed — Withdrawal by Subject | 10
Not completed — Lost to Follow-up | 2
Not completed — Lack of Efficacy | 59
Not completed — Other | 13

BASELINE CHARACTERISTICS:
Population: Intention to Treat (ITT) population: all participants who had received at least one dose of study drug and had data for at least one post-baseline assessment of any effectiveness measurement [up to and including Week 26] while receiving treatment with adalimumab.
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 461
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.8 (13.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 206
  Male | 255

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Short Inflammatory Bowel Disease Questionnaire (SIBDQ): Total Score
Description: The SIBDQ is a disease-specific health-related quality of life (HRQOL) questionnaire, able to detect and define meaningful clinical changes in inflammatory bowel disease (IBD) participants by measuring physical, social and emotional status. The SIBDQ consists of 10 questions; each question is scored on a scale from 1 (poor QOL) to 7 (optimum QOL). A higher score indicates a better health-related quality of life. Total scores range from 10 (poor QoL) to 70 (good QoL).
Time Frame: Week 0 (baseline) and Week 26
Population: All participants in the ITT population with evaluable data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 460
units on a scale | 17.4 (14.48)
Statistical Analysis 1: Comparison: Participants Receiving Adalimumab; Hypothesis testing for the first ranked primary outcome was performed in a hierarchical order using the two-sided paired t-test for mean change equal to zero; Test type: Superiority or Other; p < 0.001, paired t-test, 2 sided; Mean Difference (Final Values) = 17.40, 95% CI 2-sided [16.08 to 18.73]

2. Primary Outcome: Mean Change From the 6 Months Prior to Treatment With Adalimumab to the 6 Months After Beginning Treatment With Adalimumab in Costs of UC-related Medical Care Excluding Adalimumab Costs
Description: Medical care costs included, but were not limited to: surgical procedures, hospitalizations, bed days in hospital, unscheduled physician consultations, emergency room visits, unscheduled examination appointments, radiology appointments, endoscopy appointments and medications.
Time Frame: 6 months prior to treatment start (Week 0 [baseline]) and 6 months after treatment start (total 12 months)
Population: All participants in the ITT population with evaluable data.
Measure: Mean (Standard Deviation); unit: Pound Sterling (GBP)
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 461
Pound Sterling (GBP) | -1383.8 (2213.06)
Statistical Analysis 1: Comparison: Participants Receiving Adalimumab; Hypothesis testing for the second ranked primary outcome was performed in a hierarchical order using the two-sided paired t-test for mean change equal to zero; Test type: Superiority or Other; p < 0.001, Paired t-test, 2 sided; Mean Difference (Net) = -1383.81, 95% CI 2-sided [-1586.36 to -1181.26]

3. Secondary Outcome: Mean Change From the 6 Months Prior to Treatment With Adalimumab to the 6 Months After Beginning Treatment With Adalimumab in Total All-cause Direct Health Care Costs (Excluding Adalimumab Costs)
Description: as for outcome 2
Time Frame: 6 months prior to treatment start (Week 0 [baseline]) and 6 months after treatment start (total 12 months)
Population: All participants in the ITT population with evaluable data.
Measure: Mean (Standard Deviation); unit: Pound Sterling (GBP)
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 461
Pound Sterling (GBP) | -1297.8 (2888.89)
Statistical Analysis 1: Comparison: Participants Receiving Adalimumab; Test type: Superiority or Other; p < 0.001, Paired t-test, 2 sided; Mean Difference (Net) = -1297.77, 95% CI 2-sided [-1562.17 to -1033.36]

4. Secondary Outcome: Mean Change From the 6 Months Prior to Treatment With Adalimumab to the 6 Months After Beginning Treatment With Adalimumab in UC-related Direct and Indirect Health Care Costs
Description: UC-related direct and indirect health care costs included, but were not limited to: surgical procedures, hospitalizations, bed days in hospital, unscheduled physician consultations, emergency room visits, unscheduled examination appointments, radiology appointments, endoscopy appointments, medications and indirect costs based on WPAI.
Time Frame: 6 months prior to treatment start (Week 0 [baseline]) and 6 months after treatment start (total 12 months)
Population: All participants in the ITT population with evaluable data.
Measure: Mean (Standard Deviation); unit: Pound Sterling (GBP)
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 461
Pound Sterling (GBP) | -4308.3 (7394.75)
Statistical Analysis 1: Comparison: Participants Receiving Adalimumab; Test type: Superiority or Other; p < 0.001, Paired t-test, 2 sided; Mean Difference (Net) = -4308.32, 95% CI 2-sided [-4985.13 to -3631.51]

5. Secondary Outcome: Mean Change From the 6 Months Prior to Treatment With Adalimumab to the 6 Months After Beginning Treatment With Adalimumab in UC-related and All-cause Hospitalization
Description: Hospitalization was defined as number of bed days in hospital as determined from the health care utilization information.
Time Frame: 6 months prior to treatment start (Week 0 [baseline]) and 6 months after treatment start (total 12 months)
Population: All participants in the ITT population with evaluable data.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 158
Days | -7.3 (16.06)
Statistical Analysis 1: Comparison: Participants Receiving Adalimumab; Test type: Superiority or Other; p < 0.001, Paired t-test, 2 sided; Mean Difference (Net) = -7.3, 95% CI 2-sided [-9.83 to -4.78]

6. Secondary Outcome: Mean Change From Baseline in Participant's Satisfaction Using Treatment Satisfaction Questionnaire for Medication (TSQM)
Description: TSQM is a questionnaire to be completed by the participants to determine their satisfaction of the medications for ulcerative colitis including the study drug. The TSQM is a 14-item subject-rated scale that evaluates the effectiveness, side effects, convenience, and global satisfaction of the medication over the past 2-3 weeks. Each of the 14 questions are scored from 1 (worst) to 7 points (best); and each of the domains are scored from 0 (less satisfaction) to 100 (better satisfaction). N = participants with evaluable baseline and post-baseline data.
Time Frame: Week 0 (baseline) and Week 26
Population: All participants in the ITT population with evaluable data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 452
units on a scale
  Effectiveness (N=452) | 24.4 (31.09)
  Side Effects (N=449) | 18.9 (38.06)
  Convenience (N=451) | 6.2 (24.87)
  Global Satisfaction (N=449) | 22.6 (32.84)
Statistical Analysis 1: Comparison: Participants Receiving Adalimumab; Statistical analysis for Treatment Satisfaction Questionnaire for Medication (TSQM) Effectiveness; Test type: Superiority or Other; p < 0.001, Paired t-test, 2 sided; Mean Difference (Final Values) = 24.37, 95% CI 2-sided [21.50 to 27.25]
Statistical Analysis 2: Comparison: Participants Receiving Adalimumab; Statistical analysis for Treatment Satisfaction Questionnaire for Medication (TSQM) Side Effects; Test type: Superiority or Other; p < 0.001, Paired t-test, 2 sided; Mean Difference (Final Values) = 18.95, 95% CI 2-sided [15.42 to 22.48]
Statistical Analysis 3: Comparison: Participants Receiving Adalimumab; Statistical analysis for Treatment Satisfaction Questionnaire for Medication (TSQM) Convenience; Test type: Superiority or Other; p < 0.001, Paired t-test, 2 sided); Mean Difference (Final Values) = 6.20, 95% CI 2-sided [3.89 to 8.50]
Statistical Analysis 4: Comparison: Participants Receiving Adalimumab; Statistical analysis for Treatment Satisfaction Questionnaire for Medication (TSQM) Global Satisfaction; Test type: Superiority or Other; p < 0.001, Paired t-test, 2 sided; Mean Difference (Final Values) = 22.60, 95% CI 2-sided [19.55 to 25.64]

7. Secondary Outcome: Mean Change From the 6 Months Prior to Treatment With Adalimumab to the 6 Months After Beginning Treatment With Adalimumab in UC-related Outpatient Utilization, Including Emergency Department Visits, Unscheduled Consultation, Exam Procedures
Description: UC-related outpatient utilization was determined from the health care utilization information. Outpatient utilization was the number of procedures/surgeries performed during outpatient visits. Participants without any outpatient utilization were excluded.
Time Frame: 6 months prior to treatment start (Week 0 [baseline]) and 6 months after treatment start (total 12 months)
Population: All participants in the ITT population with evaluable data.
Measure: Mean (Standard Deviation); unit: Procedures/ Surgeries
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 453
Procedures/ Surgeries
  Overall | -4.8 (6.25)
  During emergency department visits | 0.0 (1.09)
  During primary care doctor visits | -0.9 (2.82)
Statistical Analysis 1: Comparison: Participants Receiving Adalimumab; Statistical analysis for overall UC-related outpatient utilization; Test type: Superiority or Other; p < 0.001, Paired t-test, 2 sided; Mean Difference (Net) = -4.85, 95% CI 2-sided [-5.42 to -4.27]
Statistical Analysis 2: Comparison: Participants Receiving Adalimumab; Statistical analysis for overall UC-related outpatient utilization during emergency department visits; Test type: Superiority or Other; p = 0.830, Paired t-test, 2 sided; Mean Difference (Net) = -0.01, 95% CI 2-sided [-0.11 to 0.09]
Statistical Analysis 3: Comparison: Participants Receiving Adalimumab; Statistical analysis for overall UC-related outpatient utilization during primary care doctor visits; Test type: Superiority or Other; p < 0.001, Paired t-test, 2 sided; Mean Difference (Net) = -0.92, 95% CI 2-sided [-1.18 to -0.66]

8. Secondary Outcome: Percentage of Participants With Absence of Blood in Stool
Description: Participants with absence of blood in stool were reported.
Time Frame: Week 26
Population: All participants in the ITT population with evaluable data.
Measure: Number; unit: percentage of participants
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 461
percentage of participants | 56.6
Statistical Analysis 1: Comparison: Participants Receiving Adalimumab; Statistical analysis for percentage of participants with absence of blood in stool from week 0 to week 26; Test type: Superiority or Other; p < 0.001, McNemar

9. Secondary Outcome: Mean Change From Baseline in Short Inflammatory Bowel Disease Questionnaire (SIBDQ): Total Score Over Time
Description: The SIBDQ is a disease-specific health-related quality of life (HRQoL) questionnaire, used to detect changes in inflammatory bowel disease (IBD) participants by measuring physical, social and emotional status. The SIBDQ consists of 10 questions, each question is scored on a scale from 1 (poor QoL) to 7 (good QoL). A higher score indicates a better health-related quality of life. Total scores range from 10 (poor QoL) to 70 (good QoL). N = participants with evaluable baseline and post-baseline data.
Time Frame: Week 0 (baseline), Week 2, Week 8, Week 18, and Week 26
Population: All participants in the ITT population with evaluable data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 460
units on a scale
  Week 2 (N=457) | 11.1 (9.81)
  Week 8 (N=459) | 15.4 (12.83)
  Week 18 (N=459) | 14.8 (13.06)
  Week 26 (N=460) | 17.4 (14.48)
Statistical Analysis 1: Comparison: Participants Receiving Adalimumab; Statistical analysis for mean change in SIBDQ: Total Score from week 0 to week 2; Test type: Superiority or Other; p < 0.001, Paired t-test, 2 sided; Mean Difference (Final Values) = 11.11, 95% CI 2-sided [10.21 to 12.02]
Statistical Analysis 2: Comparison: Participants Receiving Adalimumab; Statistical analysis for mean change in SIBDQ: Total Score from week 0 to week 8; Test type: Superiority or Other; p < 0.001, Paired t-test, 2 sided; Mean Difference (Final Values) = 15.38, 95% CI 2-sided [14.20 to 16.56]
Statistical Analysis 3: Comparison: Participants Receiving Adalimumab; Statistical analysis for mean change in SIBDQ: Total Score from week 0 to week 18. Efficacy assessments were not specified at week 18; missing data at week 18 were imputed using last observation carried forward (LOCF); Test type: Superiority or Other; p < 0.001, Paired t-test, 2 sided; Mean Difference (Final Values) = 14.77, 95% CI 2-sided [13.57 to 15.96]
Statistical Analysis 4: Comparison: Participants Receiving Adalimumab; Statistical analysis for mean change in SIBDQ: Total Score from week 0 to week 26; Test type: Superiority or Other; p < 0.001, Paired t-test, 2 sided; Mean Difference (Final Values) = 17.40, 95% CI 2-sided [16.08 to 18.73]

10. Secondary Outcome: Mean Change From Baseline in Physician's Global Assessment (PGA)
Description: The Physician's Global Assessment was used to measure the participant's disease activity. The physician considered the participant's reported information such as number of stools, rectal bleeding, abdominal discomfort, and functional assessment during the previous day prior to the visit, and other observations such as physical findings, and the participant's performance status at the time of the visit. Based on the above information the investigator made an overall assessment of participant's current severity of UC using the ordinal scale from 0 (normal) to 3 (severe disease).
Time Frame: Week 0 (baseline), Week 2, Week 8, Week 18, and Week 26
Population: All participants in the ITT population with evaluable data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 461
units on a scale
  Week 2 | -0.6 (0.69)
  Week 8 | -1.1 (0.85)
  Week 18 | -0.9 (0.95)
  Week 26 | -1.1 (0.97)
Statistical Analysis 1: Comparison: Participants Receiving Adalimumab; Statistical analysis for mean change in PGA from week 0 to week 2; Test type: Superiority or Other; p < 0.001, Paired t-test, 2 sided; Mean Difference (Final Values) = -0.63, 95% CI 2-sided [-0.69 to -0.57]
Statistical Analysis 2: Comparison: Participants Receiving Adalimumab; Statistical analysis for mean change in PGA from week 0 to week 8; Test type: Superiority or Other; p < 0.001, Paired t-test, 2 sided; Mean Difference (Final Values) = -1.08, 95% CI 2-sided [-1.16 to -1.00]
Statistical Analysis 3: Comparison: Participants Receiving Adalimumab; Statistical analysis for mean change in PGA from week 0 to week 18. Efficacy assessments were not specified at week 18; missing data at week 18 were imputed using LOCF; Test type: Superiority or Other; p < 0.001, Paired t-test, 2 sided; Mean Difference (Final Values) = -0.86, 95% CI 2-sided [-0.95 to -0.77]
Statistical Analysis 4: Comparison: Participants Receiving Adalimumab; Statistical analysis for mean change in PGA from week 0 to week 26; Test type: Superiority or Other; p < 0.001, Paired t-test, 2 sided; Mean Difference (Final Values) = -1.15, 95% CI 2-sided [-1.23 to -1.06]

11. Secondary Outcome: Mean Change From Baseline in Total Simple Clinical Colitis Activity Index (SCCAI)
Description: The SCCAI measures disease activity as assessed by the investigator and includes the following 6 items: bowel frequency (day), bowel frequency (night), urgency of defecation, blood in stool, general well-being and extra colonic features. The score ranges from 0 (best) to 19 points (worst).
Time Frame: Week 0 (baseline), Week 2, Week 8, Week 18, and Week 26
Population: All participants in the ITT population with evaluable data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 461
units on a scale
  Week 2 | -3.2 (2.55)
  Week 8 | -4.1 (3.33)
  Week 18 | -3.0 (3.79)
  Week 26 | -4.1 (3.88)
Statistical Analysis 1: Comparison: Participants Receiving Adalimumab; Statistical analysis for mean change in total SCCAI from week 0 to week 2; Test type: Superiority or Other; p < 0.001, Paired t-test, 2 sided; Mean Difference (Final Values) = -3.22, 95% CI 2-sided [-3.46 to -2.99]
Statistical Analysis 2: Comparison: Participants Receiving Adalimumab; Statistical analysis for mean change in total SCCAI from week 0 to week 8; Test type: Superiority or Other; p < 0.001, Paired t-test, 2 sided; Mean Difference (Final Values) = -4.06, 95% CI 2-sided [-4.37 to -3.76]
Statistical Analysis 3: Comparison: Participants Receiving Adalimumab; Statistical analysis for mean change in total SCCAI from week 0 to week 18. Efficacy assessments were not specified at week 18; missing data at week 18 were imputed using LOCF; Test type: Superiority or Other; p < 0.001, Paired t-test, 2 sided; Mean Difference (Final Values) = -3.01, 95% CI 2-sided [-3.36 to -2.66]
Statistical Analysis 4: Comparison: Participants Receiving Adalimumab; Statistical analysis for mean change in total SCCAI from week 0 to week 26; Test type: Superiority or Other; p < 0.001, Paired t-test, 2 sided; Mean Difference (Final Values) = -4.07, 95% CI 2-sided [-4.43 to -3.72]

12. Secondary Outcome: Mean Change From Baseline in European Quality of Life - 5 Dimensions - 5 Level (EQ-5D-5L) Total Score
Description: EQ-5D-5L Total Score provides a descriptive profile of health status. It comprises of 5 dimensions of health (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) to describe the subject's current health state. Each dimension comprises 5 levels with corresponding numeric scores ranging from 1 (no problems) through 5 (extreme problems). A unique EQ-5D-5L health state was defined by combining the numeric level scores for each of the 5 dimensions and the total score ranges from -0.594 to 1, with higher scores representing a better health state. An increase in the EQ-5D-5L total score indicates improvement. N = participants with evaluable baseline and post-baseline data.
Time Frame: Week 0 (baseline), Week 2, Week 8, Week 18, and Week 26
Population: All participants in the ITT population with evaluable data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 454
units on a scale
  Week 2 (N=452) | 0.1 (0.18)
  Week 8 (N=454) | 0.1 (0.21)
  Week 18 (N=454) | 0.1 (0.22)
  Week 26 (N=454) | 0.1 (0.23)
Statistical Analysis 1: Comparison: Participants Receiving Adalimumab; Statistical analysis for mean change in total EQ-5D-5L total score from week 0 to week 2; Test type: Superiority or Other; p < 0.001, Paired t-test, 2 sided; Mean Difference (Final Values) = 0.10, 95% CI 2-sided [0.08 to 0.11]
Statistical Analysis 2: Comparison: Participants Receiving Adalimumab; Statistical analysis for mean change in total EQ-5D-5L total score from week 0 to week 8; Test type: Superiority or Other; p < 0.001, Paired t-test, 2 sided; Mean Difference (Final Values) = 0.13, 95% CI 2-sided [0.11 to 0.15]
Statistical Analysis 3: Comparison: Participants Receiving Adalimumab; Statistical analysis for mean change in total EQ-5D-5L total score from week 0 to week 18. Efficacy assessments were not specified at week 18; missing data at week 18 were imputed using LOCF; Test type: Superiority or Other; p < 0.001, Paired t-test, 2 sided; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [0.10 to 0.14]
Statistical Analysis 4: Comparison: Participants Receiving Adalimumab; Statistical analysis for mean change in total EQ-5D-5L total score from week 0 to week 26; Test type: Superiority or Other; p < 0.001, Paired t-test, 2 sided; Mean Difference (Final Values) = 0.14, 95% CI 2-sided [0.12 to 0.17]

13. Secondary Outcome: Mean Change From Baseline in Work Productivity and Activity Impairment Questionnaire: Specific Health Problem (WPAI-SHP): Percentage of Work Time Missed
Description: WPAI-SHP is a questionnaire used to assess the effect of the participant's health problems on their ability to work and perform regular activities. A higher score indicates an increased impairment. A positive value of change indicates an increased impairment of work productivity and the limitation of activities of daily life, while a negative value indicates an improvement. The percentage of work time missed data was applicable to employed participants only. N = participants with evaluable baseline and post-baseline data.
Time Frame: Week 0 (baseline), Week 2, Week 8, Week 18, and Week 26
Population: All participants in the ITT population with evaluable data.
Measure: Mean (Standard Deviation); unit: percentage of work time missed
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 227
percentage of work time missed
  Week 2 (N=214) | -8.6 (25.55)
  Week 8 (N=227) | -12.2 (30.97)
  Week 18 (N=225) | -11.6 (32.04)
  Week 26 (N=223) | -11.4 (30.85)
Statistical Analysis 1: Comparison: Participants Receiving Adalimumab; Statistical analysis for mean change in WPAI-SHP: percentage of work time missed from week 0 to week 2; Test type: Superiority or Other; p < 0.001, Paired t-test, 2 sided; Mean Difference (Final Values) = -8.62, 95% CI 2-sided [-12.07 to -5.18]
Statistical Analysis 2: Comparison: Participants Receiving Adalimumab; Statistical analysis for mean change in WPAI-SHP: percentage of work time missed from week 0 to week 8; Test type: Superiority or Other; p < 0.001, Paired t-test, 2 sided; Mean Difference (Final Values) = -12.22, 95% CI 2-sided [-16.27 to -8.16]
Statistical Analysis 3: Comparison: Participants Receiving Adalimumab; Statistical analysis for mean change in WPAI-SHP: percentage of work time missed from week 0 to week 18. Efficacy assessments were not specified at week 18; missing data at week 18 were imputed using last observation carried forward (LOCF); Test type: Superiority or Other; p < 0.001, Paired t-test, 2 sided; Mean Difference (Final Values) = -11.61, 95% CI 2-sided [-15.82 to -7.40]
Statistical Analysis 4: Comparison: Participants Receiving Adalimumab; Statistical analysis for mean change in WPAI-SHP: percentage of work time missed from week 0 to week 26; Test type: Superiority or Other; p < 0.001, Paired t-test, 2 sided; Mean Difference (Final Values) = -11.43, 95% CI 2-sided [-15.50 to -7.35]

14. Secondary Outcome: Mean Change From Baseline in Work Productivity and Activity Impairment Questionnaire: Specific Health Problem (WPAI-SHP): Percentage of Impairment While Working
Description: WPAI-SHP is a questionnaire used to assess the effect of the participant's health problems on their ability to work and perform regular activities. The scores on the WPAI questionnaire are presented as percentages (multiplying the scores by 100), with 0% representing no impact on productivity and 100% representing complete impact on productivity. Change in WPAI-SHP was calculated by deducting the final score from the baseline score. A higher score indicates an increased impairment. A positive value of change indicates an increased impairment of work productivity and the limitation of activities of daily life, while a negative value indicates an improvement. The percentage of impairment while working data was applicable to employed participants only. N = participants with evaluable baseline and post-baseline data.
Time Frame: Week 0 (baseline), Week 2, Week 8, Week 18, and Week 26
Population: All participants in the ITT population with evaluable data.
Measure: Mean (Standard Deviation); unit: percentage of impairment while working
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 234
percentage of impairment while working
  Week 2 (N=221) | -16.6 (25.94)
  Week 8 (N=234) | -22.9 (30.91)
  Week 18 (N=232) | -21.7 (30.98)
  Week 26 (N=229) | -24.5 (29.78)
Statistical Analysis 1: Comparison: Participants Receiving Adalimumab; Statistical analysis for mean change in WPAI-SHP: percentage of impairment while working from week 0 to week 2; Test type: Superiority or Other; p < 0.001, Paired t-test, 2 sided; Mean Difference (Final Values) = -16.56, 95% CI 2-sided [-20.00 to -13.12]
Statistical Analysis 2: Comparison: Participants Receiving Adalimumab; Statistical analysis for mean change in WPAI-SHP: percentage of impairment while working from week 0 to week 8; Test type: Superiority or Other; p < 0.001, Paired t-test, 2 sided; Mean Difference (Final Values) = -22.95, 95% CI 2-sided [-26.93 to -18.97]
Statistical Analysis 3: Comparison: Participants Receiving Adalimumab; Statistical analysis for mean change in WPAI-SHP: percentage of impairment while working from week 0 to week 18. Efficacy assessments were not specified at week 18; missing data at week 18 were imputed using last observation carried forward (LOCF); Test type: Superiority or Other; p < 0.001, Paired t-test, 2 sided; Mean Difference (Final Values) = -21.68, 95% CI 2-sided [-25.69 to -17.67]
Statistical Analysis 4: Comparison: Participants Receiving Adalimumab; Statistical analysis for mean change in WPAI-SHP: percentage of impairment while working from week 0 to week 26; Test type: Superiority or Other; p < 0.001, Paired t-test, 2 sided; Mean Difference (Final Values) = -24.45, 95% CI 2-sided [-28.33 to -20.58]

15. Secondary Outcome: Mean Change From Baseline in Work Productivity and Activity Impairment Questionnaire: Specific Health Problem (WPAI-SHP): Overall Work Impairment Percentage
Description: WPAI-SHP is a questionnaire used to assess the effect of the participant's health problems on their ability to work and perform regular activities. The scores on the WPAI questionnaire are presented as percentages (multiplying the scores by 100), with 0% representing no impact on productivity and 100% representing complete impact on productivity. Change in WPAI-SHP was calculated by deducting the final score from the baseline score. A higher score indicates an increased impairment. A positive value of change indicates an increased impairment of work productivity and the limitation of activities of daily life, while a negative value indicates an improvement. The overall work impairment data was applicable to employed participants only. N = participants with evaluable baseline and post-baseline data.
Time Frame: Week 0 (baseline), Week 2, Week 8, Week 18, and Week 26
Population: All participants in the ITT population with evaluable data.
Measure: Mean (Standard Deviation); unit: percentage of overall work impairment
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 225
percentage of overall work impairment
  Week 2 (N= 211) | -18.3 (27.72)
  Week 8 (N= 225) | -26.5 (34.56)
  Week 18 (N= 223) | -25.3 (35.10)
  Week 26 (N= 221) | -29.2 (32.32)
Statistical Analysis 1: Comparison: Participants Receiving Adalimumab; Statistical analysis for mean change in WPAI-SHP: overall work impairment percentage from week 0 to week 2; Test type: Superiority or Other; p < 0.001, Paired t-test, 2 sided; Mean Difference (Final Values) = -18.34, 95% CI 2-sided [-22.10 to -14.57]
Statistical Analysis 2: Comparison: Participants Receiving Adalimumab; Statistical analysis for mean change in WPAI-SHP: overall work impairment percentage from week 0 to week 8; Test type: Superiority or Other; p < 0.001, Paired t-test, 2 sided; Mean Difference (Final Values) = -26.54, 95% CI 2-sided [-31.08 to -22.00]
Statistical Analysis 3: Comparison: Participants Receiving Adalimumab; Statistical analysis for mean change in WPAI-SHP: overall work impairment percentage from week 0 to week 18. Efficacy assessments were not specified at week 18; missing data at week 18 were imputed using LOCF; Test type: Superiority or Other; p < 0.001, Paired t-test, 2 sided; Mean Difference (Final Values) = -25.33, 95% CI 2-sided [-29.97 to -20.70]
Statistical Analysis 4: Comparison: Participants Receiving Adalimumab; Statistical analysis for mean change in WPAI-SHP: overall work impairment percentage from week 0 to week 26; Test type: Superiority or Other; p < 0.001, Paired t-test, 2 sided; Mean Difference (Final Values) = -29.22, 95% CI 2-sided [-33.50 to -24.93]

16. Secondary Outcome: Mean Change From Baseline in Work Productivity and Activity Impairment Questionnaire: Specific Health Problem (WPAI-SHP): Percentage of Activity Impairment
Description: WPAI-SHP is a questionnaire used to assess the effect of the participant's health problems on their ability to work and perform regular activities. The scores on the WPAI questionnaire are presented as percentages (multiplying the scores by 100), with 0% representing no impact on productivity and 100% representing complete impact on productivity. Change in WPAI-SHP was calculated by deducting the final score from the baseline score. A higher score indicates an increased impairment. A positive value of change indicates an increased impairment of work productivity and the limitation of activities of daily life, while a negative value indicates an improvement. N = participants with evaluable baseline and post-baseline data.
Time Frame: Week 0 (baseline), Week 2, Week 8, Week 18, and Week 26
Population: All participants in the ITT population with evaluable data.
Measure: Mean (Standard Deviation); unit: percentage of activity impairment
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 446
percentage of activity impairment
  Week 2 (N=435) | -18.2 (24.55)
  Week 8 (N=446) | -25.4 (30.84)
  Week 18 (N=446) | -24.4 (31.35)
  Week 26 (N-446) | -27.2 (32.83)
Statistical Analysis 1: Comparison: Participants Receiving Adalimumab; Statistical analysis for mean change in WPAI-SHP: percentage of activity impairment from week 0 to week 2; Test type: Superiority or Other; p < 0.001, Paired t-test, 2 sided; Mean Difference (Final Values) = -18.16, 95% CI 2-sided [-20.47 to -15.85]
Statistical Analysis 2: Comparison: Participants Receiving Adalimumab; Statistical analysis for mean change in WPAI-SHP: percentage of activity impairment from week 0 to week 8; Test type: Superiority or Other; p < 0.001, Paired t-test, 2 sided; Mean Difference (Final Values) = -25.43, 95% CI 2-sided [-28.30 to -22.56]
Statistical Analysis 3: Comparison: Participants Receiving Adalimumab; Statistical analysis for mean change in WPAI-SHP: percentage of activity impairment from week 0 to week 18. Efficacy assessments were not specified at week 18; missing data at week 18 were imputed using last observation carried forward (LOCF); Test type: Superiority or Other; p < 0.001, Paired t-test, 2 sided; Mean Difference (Final Values) = -24.42, 95% CI 2-sided [-27.33 to -21.50]
Statistical Analysis 4: Comparison: Participants Receiving Adalimumab; Statistical analysis for mean change in WPAI-SHP: percentage of activity impairment from week 0 to week 26; Test type: Superiority or Other; p < 0.001, Paired t-test, 2 sided; Mean Difference (Final Values) = -27.22, 95% CI 2-sided [-30.28 to -24.16]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from the time of study drug administration to 70 days after last dose of study drug (up to 36 weeks).
Description: Serious Adverse Events were also collected from the time that informed consent was obtained until 70 days after last dose (up to 39 weeks).
Arm/Group | PARTICIPANTS RECEIVING ADALIMUMAB
Serious Adverse Events (participants affected / at risk) | 67/463
Other Adverse Events (participants affected / at risk) | 178/463
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PARTICIPANTS RECEIVING ADALIMUMAB (N=463)
ANAEMIA (Blood and lymphatic system disorders) | 2
PANCYTOPENIA (Blood and lymphatic system disorders) | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1
SILENT MYOCARDIAL INFARCTION (Cardiac disorders) | 1
HYPERTHYROIDISM (Endocrine disorders) | 1
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 1
COLITIS ULCERATIVE (Gastrointestinal disorders) | 41
DIARRHOEA (Gastrointestinal disorders) | 1
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1
MEGACOLON (Gastrointestinal disorders) | 1
ACCIDENTAL DEATH (General disorders) | 1
ASTHENIA (General disorders) | 1
APPENDICITIS (Infections and infestations) | 1
CELLULITIS (Infections and infestations) | 1
CYTOMEGALOVIRUS INFECTION (Infections and infestations) | 1
GASTROENTERITIS (Infections and infestations) | 1
HERPES ZOSTER (Infections and infestations) | 1
OSTEOMYELITIS (Infections and infestations) | 1
OTITIS MEDIA (Infections and infestations) | 1
PYELONEPHRITIS (Infections and infestations) | 1
RECTAL ABSCESS (Infections and infestations) | 1
SINUSITIS (Infections and infestations) | 1
WOUND SEPSIS (Infections and infestations) | 1
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 1
PNEUMOTHORAX TRAUMATIC (Injury, poisoning and procedural complications) | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1
OSTEITIS (Musculoskeletal and connective tissue disorders) | 1
MALIGNANT MELANOMA OF EYELID (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
TESTICULAR SEMINOMA (PURE) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 1
DIZZINESS (Nervous system disorders) | 1
INTRACRANIAL VENOUS SINUS THROMBOSIS (Nervous system disorders) | 1
FOETAL DEATH (Pregnancy, puerperium and perinatal conditions) | 1
FOETAL DISTRESS SYNDROME (Pregnancy, puerperium and perinatal conditions) | 1
DEPRESSION (Psychiatric disorders) | 1
DERMATOSIS (Skin and subcutaneous tissue disorders) | 1
PRURITUS GENERALISED (Skin and subcutaneous tissue disorders) | 1
ABORTION INDUCED (Surgical and medical procedures) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PARTICIPANTS RECEIVING ADALIMUMAB (N=463)
COLITIS ULCERATIVE (Gastrointestinal disorders) | 61
NAUSEA (Gastrointestinal disorders) | 29
NASOPHARYNGITIS (Infections and infestations) | 37
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 33
HEADACHE (Nervous system disorders) | 60
COUGH (Respiratory, thoracic and mediastinal disorders) | 27
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.